CLINICAL TRIAL: NCT00434681
Title: Multicentre, Open, Non-Comparative Study of the Acceptability and Safety of Paracetamol Oral Paediatric Suspension at 4.8%.
Brief Title: Paracetamol Oral Paediatric Suspension at 4.8% : Study of Acceptability and Safety.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: PARAC_L_00859
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Last update posted 2008-07-21 (Estimated); Status verified 2008-07

CONDITIONS: Fever; Pain
MeSH Terms: conditions — Fever; Pain | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: paracetamol 4.8% paediatric oral suspension

SUMMARY:
Evaluate the acceptability over 24 hours of a new paracetamol formulation 4.8% paediatric oral suspension in children weighing between 3 and 26 kg including limits

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Main criteria are listed hereafter :

Inclusion Criteria:

* Children of both sexes weighing between 3 and 26 kg including limits.
* With a fever and/or painful episode justifying a paracetamol treatment for a minimum duration of 24 hours.
* Likely to be followed throughout the entire study period in out-patient.
* For whom the informed consent has been signed by the parents or legal guardian and by the child if old enough (see chapter 12.3).

Exclusion Criteria:

* Presenting digestive disorders, vomiting.
* Presenting a hypersensitivity to paracetamol or one of the ingredients of the study product
* Presenting a hepatocellular failure.
* Presenting a fructose intolerance.
* Presenting a serious concomitant disease, such as cancer, immune deficiency or a serious renal, hepatic cardiac, neurological, psychiatric or metabolic disease.
* Presenting a history of significant biological anomalies.
* Treated with Kayexalate® (sodium polystyrene sulphonate)
* Not covered by a social security regime.
* Whose parents are incapable of understanding
* Who cannot come back to the consultation for the final evaluation and/or submit to the study constraints.
* Who participated in another clinical study in the 30 days prior to inclusion.
* Is a relation of the investigator.

Ages: 1 Day to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48
Dates: Start 2006-10; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Acceptability data: Overall evaluation of the treatment by the child's parents or the minder, measured using a semi-quantitative scale with 4 levels (very acceptable, acceptable, indifferent, refusal), for 24 hours (4 evaluations at 6 hour intervals).
Safety data : Events reported by the child, parents or legal guardian during visit 2 ; events compiled in the child's diary ; events recorded by the investigator during Visit 2

SECONDARY OUTCOMES:
Acceptability data: Overall evaluation of the child (from 3 years), using a Hedonic Visual Scale during the last administration prior to Visit V2.

CONTACTS AND LOCATIONS:
Overall Officials: Monique COUDERC, Dr, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France